CLINICAL TRIAL: NCT02525341
Title: Yoga Versus Aerobic and Strengthening Exercises for Managing Knee Osteoarthritis
Brief Title: Yoga Versus Exercises for Managing OA
Acronym: YEMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1212M25141
Record Dates: First submitted 2015-07-20; First posted 2015-08-17 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Knee Osteoarthritis
Keywords: Yoga; exercises; knee osteoarthritis; older adults
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity | interventions — Yoga

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Yoga Group (Experimental): Participants in the yoga group received a total of eight weekly 45 minute yoga classes. A sequence of 8 - 10 core yoga poses, breathing and relaxation techniques were practiced in each yoga class, and 2 - 3 new poses were introduced progressively in each of the yoga session. Props such as blocks, blankets, belts, mats, and chairs were used during the session. Handouts were provided for participants to practice the yoga program for additional 30 minutes a day, 4 days a week at home.
  Interventions: Other: Hatha yoga
- Aerobic and Strengthening Exercise Group (Active Comparator): Participants in the exercise group received a total of eight weekly 45 minute exercise classes. A 15 minute of gentle aerobic exercise and a 30 minute of strengthening program that includes both isometric (without moving the joints) and isotonic (moving the joints) exercises of the lower extremities were taught to the participants. Handouts were provided for participants to practice the program at home for 30 minutes a day, 3 days a week (on non-consecutive days).
  Interventions: Other: Aerobic and strengthening exercises
- General education (Active Comparator): Participants in this group received a one-time OA educational brochures from the Arthritis Foundation including topics focusing on the disease process, diet and exercise and OA management education. Participants were instructed not to begin any new exercise programs during the study period.
  Interventions: Other: General education

INTERVENTIONS:
Other: Hatha yoga — A sequence of 8 - 10 core yoga poses, breathing and relaxation techniques were practiced in each yoga class, and 2 - 3 new poses were introduced progressively in each of the yoga session. Props such as blocks, blankets, belts, mats, and chairs were used during the session.
  Other Names: Yoga
  Arms: Yoga Group
Other: Aerobic and strengthening exercises — A 15 minute of gentle aerobic exercise and a 30 minute of strengthening program that includes both isometric (without moving the joints) and isotonic (moving the joints) exercises of the lower extremities were taught to the participants.
  Arms: Aerobic and Strengthening Exercise Group
Other: General education — One-time Arthritis Foundation educational brochures focusing on the disease process, diet and exercise and OA management education were given.
  Arms: General education

SUMMARY:
The purpose of the study is to examine the short and long term effects of Hatha yoga compared to the current recommended exercise program in promoting physical function, alleviating osteoarthritis (OA)-related symptoms, fear of falling, and improving mood, spiritual health, physical activity level, and quality of life in older adults with knee OA, and to determine the effect sizes for use in power calculations to design a larger efficacy clinical trial.

DETAILED DESCRIPTION:
The specific aims of this pilot project are to:

Aim 1: Examine the short and long term effect of participation in an 8-week intervention of Hatha yoga (HY) on pain, stiffness, physical function of the lower extremities, physical activity, mood, fear of falling, spiritual health, and quality of life in older women with knee OA, compared with the effect in those older adults who participated in aerobic/strengthening exercise (AE) or received general OA education (GE).

Aim 2: Describe the adherence rate (class and home practices) and exercise acceptability of the HY and AE programs.

A randomized controlled trial design with three groups were used: 1) A Hatha yoga (HY) intervention group, 2) an aerobic and local muscle strengthening exercise (AE) control group, and 3) a general OA education (GE) true control group. Both yoga and exercise groups involved group and home practice sessions. Participants in the GE group received education on OA management after randomization. A weekly phone call were placed to them during the intervention period to reinforce OA knowledge. Data were collected from all participants at baseline, 4 weeks, and 8 weeks during the intervention, and quarterly for one year during the follow up period.

Study Endpoints

1. Primary endpoint: OA status (pain, stiffness and function) at 8 weeks.
2. Secondary endpoint: physical function of lower extremities, mood, and quality of life at 8 weeks.
3. Tertiary endpoint: Long term exercise adherence and effects on outcome measures, program acceptability, and safety.

Sample Size and Recruitment Eight-three community dwelling older adults ages 60 years - 100 years old with a diagnosis of symptomatic knee OA were recruited. Recruitment were done through conducting presentations at various senior centers; distributing press release to various community newsletters, local and senior newspapers, and through working with my co-investigators, and accessing the data base and mailing invitation letters out to patients meeting demographic and diagnostic criteria from the University of Minnesota Physician Practice.

Each weekly group based session is 45 minute in length for all groups. Participants in the yoga group were recommended to practice for additional 30 minutes four times a week at home. Participants in the A/E class were recommended to practice 3 times on non-consecutive days at home as recommended by the current physical activity guidelines for older adults. To assist participants with maintaining exercise adherence and practicing yoga and aerobic/strengthening exercises at home correctly, handouts illustrating yoga/exercise activity were distributed at the end of each class. Participants also were asked to videotape and keep a log of their exercise practice during the intervention period. Video camera were provided. Long term exercise adherence was assessing using an exercise diary. Participants were asked to keep an exercise diary during the follow up period. A focus group will be conducted at the end of the follow-up period to examine the experience of using HY or AE for managing knee OA, and factors that affect participants' HY/AE adherence.

Descriptive statistics will be used to analyze and report demographic data and feasibility/acceptability data. Inferential statistics (t-test or non-parametric equivalent such as Mann-Whitney, and chi-square test) will be used to analyze the OA symptoms, physical and psychological outcomes. The α level will be set at ≤ .05.

ELIGIBILITY:
Inclusion Criteria:

* have been diagnosed with symptomatic OA of knee for at least 6 months,
* have not practiced any form of yoga for at least 2 months; and
* not currently participating in a supervised exercise program. "Currently" is defined as not participating in a supervised exercise program more than 2 times a week at the time of second-step screening.

Exclusion Criteria:

* OA is asymptomatic,
* have moderate/severe cognitive impairment, scored less than 8 on the Short Portable Mental Status Questionnaire,
* have cardiovascular risk,
* reported symptoms of joint locking,
* instability indicated by chronic use of a knee brace, cane, walker, or wheelchair,
* corticosteroid injection in the symptomatic joint within 3 months of study entry,
* hyaluronic acid injection: hyaluronan (Hyalgan) and synthetic hylan G-F 20 (Synvisc) in the symptomatic joint within 6 months of study entry,
* history of knee surgery within the last two years, arthroscopic lavage within 6 months, or a joint replacement of the lower extremities at any point,
* self-reported significant medical comorbidities such as: 1) uncontrolled high blood pressure or existing heart condition; and 2) other comorbid condition with overlapping symptoms (i.e. fibromyalgia, rheumatoid arthritis),
* Individuals who have medication changes for arthritis symptoms will be permitted to remain in the trial; however, these changes will be monitored.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2013-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Osteoarthritis (OA) symptoms change | Change from baseline OA symtptoms at 8 weeks
  OA pain, stiffness and function (total score) is evaluated using the Western Ontario and McMaster Universities OA (WOMAC) index scale.
Knee OA pain change | Change from baseline pain score at 8 weeks
  Visual Analog Scale
Knee OA pain change | Change from baseline number of medication used per day for OA pain at 8 weeks
  Number of pain medication used per day for OA pain

SECONDARY OUTCOMES:
Physical function | 4 and 8 weeks
  The Short Physical Performance Battery, which includes repeated chair stands, balance and 8 foot walk tests, is used to evaluate participants' physical function of lower extremities.
Gait speed | 4 and 8 weeks
  50 foot walk is used to measure gait speed.
Physical activity level | 4 and 8 weeks
  Physical Activity Scale for the Elderly is used to evaluate the different physical activity levels: leisure time activity, household activity, and work-related activity.
Fear of falling | 4 and 8 weeks
  Fear of falling is evaluated using the Falls Efficacy Scale-International.
Spiritual health | 4 and 8 weeks
  Self-Transcendence Scale is used to evaluate participants' spiritual health.
Quality of life | 4 and 8 weeks
  SF 12 v2 Health Survey is used for measuring quality of life.
Mood | 4 and 8 weeks
  Hospital Anxiety and Depression Scale is used to evaluate mood.

OTHER OUTCOMES:
Feasibility - number of eligible subjects | Baseline
  Number of eligible subjects will be assessed by the total number of subjects enrolled in the study.
Feasibility - exercise adherence | 8 weeks
  Exercise adherence will be assessed base on the:
  1. Average class attendance (weekly class attendance sheet recorded by the RA)
  2. Frequency of home practice: the average number of days per week, and the average number of minutes per day (participants' weekly self-report on an exercise log sheet).
Feasibility - adverse events | 8 weeks
  RA will record any number or type of yoga related adverse events during the intervention classes. Participants will record any number or type of yoga related adverse events during their home practice on the exercise log sheet.
Feasibility - retention rate | 8 weeks
  Retention rate will be assessed by the number of participants remain in the study.
Acceptability | 8 weeks
  An investigator-developed survey using a 10 point Likert scale will be used to assess participants' self-report satisfaction with the intervention program, perceived appropriateness of the program, and intention to continue to use the intervention program.

CONTACTS AND LOCATIONS:
Overall Officials: Corjena Cheung, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheung C, Wyman JF, Bronas U, McCarthy T, Rudser K, Mathiason MA. Managing knee osteoarthritis with yoga or aerobic/strengthening exercise programs in older adults: a pilot randomized controlled trial. Rheumatol Int. 2017 Mar;37(3):389-398. doi: 10.1007/s00296-016-3620-2. Epub 2016 Dec 2. PMID 27913870